CLINICAL TRIAL: NCT04813614
Title: SMILE Study: Effectiveness and Safety of STYLAGE® M Lidocaïne for Lips' Volume Augmentation and/or Redefinition of the Outline of the Lips
Brief Title: Effectiveness and Safety of STYLAGE® M Lidocaïne for Lips' Volume Augmentation and/or Redefinition of the Outline of the Lips (SMILE)
Acronym: SMILE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Laboratoires Vivacy (Industry)
Collaborators: Eurofins (Industry); Inferential (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2021-A00089-32
Record Dates: First submitted 2021-03-22; First posted 2021-03-24 (Actual); Last update posted 2022-11-23 (Actual); Status verified 2022-11

CONDITIONS: Esthetics
Keywords: hyaluronic acid; lips; volume; outline

STUDY DESIGN:
Intervention Model Description: Prospective, double blinded, randomized, active controlled, multicenter study (post-market clinical follow-up).
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: The subjects randomized in the study will be blinded to the treatment administered by using a blindfold during injection session(s).
  All the evaluators and operators who will take part in the investigation will be different than the legally qualified clinical practitioners who will realize injections and will be blinded to the treatment administered:
  * Live blinded independent evaluators will oversee the inclusions of subjects, the follow-up of subject's tolerance and the scoring in live of the GAIS (also using the photograph taken at V1 before first injection as a reference). The same blinded independent evaluator will follow-up the same subjects over the study period as far as possible.
  * Technicians who will oversee the photographs taking.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- STYLAGE M Lidocaine (Experimental): The first injection is performed at visit 1 (V1) on Day 0 (D0). D0 is considered as the baseline. The maximum volume to be injected is 2 mL in total for lower and upper lips. The exact volume per lip will be determined by the physician/injector in order to reach optimal volume correction and/or lips' redefinition, as well as the injection technique(s) to be used. Injection is done into and/or around the lip mucosa by linear threading injection, multipoint injection, or a combination of both techniques with needle or cannula.
  One optional touch-up injection is allowed at visit 2 (V2) on Month 1 (M1), with a maximum volume to be injected of 1 mL in total for lower and upper lips. No other touch-up injection is allowed until the end of the study.
  A total maximum volume of 2.5 mL is recommended for both initial and touch-up injections combined (upper and lower lips).
  Interventions: Device: STYLAGE M Lidocaine
- Active control group (Active Comparator): The first injection is performed at visit 1 (V1) on Day 0 (D0). D0 is considered as the baseline. The maximum volume to be injected is 2 mL in total for lower and upper lips. The exact volume per lip will be determined by the physician/injector in order to reach optimal volume correction and/or lips' redefinition, as well as the injection technique(s) to be used. Injection is done into the submucosal layer of the lip by linear threading injection or serial puncture techniques injection with needle or cannula.
  One optional touch-up injection is allowed at visit 2 (V2) on Month 1 (M1), with a maximum volume to be injected of 1 mL in total for lower and upper lips. No other touch-up injection is allowed until the end of the study.
  A total maximum volume of 2.5 mL is recommended for both initial and touch-up injections combined (upper and lower lips).
  Interventions: Device: Active control group

INTERVENTIONS:
Device: STYLAGE M Lidocaine — Injection in the lips
  Arms: STYLAGE M Lidocaine
Device: Active control group — Injection in the lips
  Arms: Active control group

SUMMARY:
STYLAGE® M Lidocaine is a hyaluronic acid injectable gel CE (conformité européenne)-marketed since 2009 . It is indicated for the outline of the lips and/or for lips augmentation in lips mucosa. It is also indicated to fill skin depressions on the face. Lidocaine is intended to reduce the pain associated with the injection.

The aim of SMILE study is to demonstrate that STYLAGE® M Lidocaine is non-inferior to an active comparator that has shown its effectiveness in lips' volume augmentation and restoration in improving the aesthetic appearance of the lips evaluated by subjects.

In this study, 92 healthy volunteers between 18 and 65 years old, who expressed the wish for augmentation or restoration of the volume of the lips and/or lips' outline redefinition, confirmed by investigators at inclusion, who have given his/her informed consent and who met all the eligibility criteria, will be enrolled.

Subjects will randomly receive STYLAGE® M Lidocaïne or the active comparator (ratio 1:1) injection in the lips at first visit on Day 0. At second visit, one month after Day 0, an optional touch-up injection could be performed according to subject's and investigator's opinions and if the subject is still eligible.

Subjects will have a total of 6 visits over a 12 months follow-up period and a screening visit prior to first injection.

Proportion of subjects having a global aesthetic improvement of their lips (blinded self-evaluation), 3 months after treatment initiation will be assessed and compared between the two groups. This will also be done during the other visits (1, 6, 9 and 12 months after treatment initiation). Global aesthetic improvement according to blinded independent evaluator, subjects' satisfaction, pain during injection and safety parameters will also be assessed during the study period.

DETAILED DESCRIPTION:
This is a prospective, double blinded, randomized, active controlled, multicenter study. Subjects are randomly assigned to receive either STYLAGE® M Lidocaine or the active comparator (ratio 1:1).

Ninety two subjects between 18 and 65 years old who expressed the wish for augmentation or restoration of the volume of the lips and/or lips' outline redefinition, confirmed by investigators at inclusion, who have given his/her informed consent and who met all the eligibility criteria (especially according to the instructions for use of the devices), will be include.

After a screening visit for selection, each subject will be followed for 12 months after 1st injection at Visit 1 (on Day 0). Five follow-up visits are scheduled 1, 3, 6, 9 and 12 months after initial injection (Visits 2 to 6). At 1 month (Visit 2), an optional touch-up injection may be done (if needed).

The primary objective is to demonstrate non-inferiority of STYLAGE® M Lidocaine versus the active comparator in improving the aesthetic appearance of the lips. The comparison of effectiveness between the devices will be done according to proportion of subjects having an improvement on the 5-point Global Aesthetic Improvement Scale (GAIS) evaluated by the blinded subject on the lips (after mirror self-examination), 3 months after treatment initiation (V1). Improvement according to GAIS corresponds to one of these three categories: "Very much improved", "Much improved" or "Improved".

Secondary objectives include subjects' self-evaluation of their lips according to GAIS, at 1, 6, 9 and 12 months after treatment initiation. Global aesthetic improvement of the lips according to blinded independent evaluator, subjects' satisfaction, subjects' self-evaluation of pain during injection will also be measured and collected at each visit during the whole study period. Study products tolerance will be assessed by collection of injection site reactions after each injection session, and adverse events throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteer.
* Sex: female or male.
* Age: between 18 and 65 years.
* Subject having given freely and expressly his/her informed consent and data privacy consent.
* Subject who expressed the wish for augmentation or restoration of the volume of the lips and/or lips' outline redefinition.
* Lips requiring volume and/or lips' outline requiring redefinition according to the investigator's judgement.
* Subject with attainable expectations for lips' volume augmentation or restoration and/or outline redefinition.
* Subject willing to have photographs of the face taken.
* Subject psychologically able to understand the study related information and to give a written informed consent.
* Subject able and agreeing to follow study procedures, instructions and likely to complete all required visits.
* Subject affiliated to a health social security system.
* Female of childbearing potential should use a medically accepted contraceptive regimen since at least 12 weeks before screening visit and during all the study.
* Subject agreeing to be treated with hyaluronidase product in case of vascular complication at the injection site.

Exclusion Criteria:

* Subject who had been deprived of their freedom by administrative or legal decision or who is under guardianship.
* Subject in a social or sanitary establishment.
* For France only: subject having received 4500 euros indemnities for participation in researches involving human beings in France in the 12 previous months, including participation in the present study).
* Subject participating to another research on human beings or who is in an exclusion period of one.
* Pregnant or breastfeeding woman or planning a pregnancy during the study.
* Subject with scar(s), mole(s) or anything on the studied zones, which might interfere with the evaluation (tattoo, permanent make-up…), including lips presenting a marked asymmetry (especially when smiling) and missing front tooth or teeth.
* Subjects with severe perioral wrinkles and seeking for upper cutaneous lip or perioral rejuvenation.
* Subject suffering from a severe or progressive disease or any other pathology that may interfere with the evaluation of the study results and/or subject safety (e.g. on-going active infection).
* Subject suffering from epilepsy, impaired cardiac conduction, severely impaired hepatic function, or severe renal dysfunction.
* Subject with known history of or suffering from autoimmune disease and/or immune deficiency.
* Subject suffering from active disease such as inflammation, infection (including oral or dental localisations), tumours, inflammatory and/or infectious cutaneous disorders (herpes, acne…) on or around the lips. Subject with history of herpes is not eligible even if asymptomatic at time of inclusion.
* Subjects suffering from porphyria.
* Subject having history of allergy or anaphylactic shock including known hypersensitivity to one of the ingredient of tested devices (i.e. hyaluronic acid, lidocaine) or to any other component of the devices used in this study, to gram-positive bacterial proteins, to antiseptic solution or to amide-type local anaesthetics.
* Subject with a history of streptococcal disease, such as acute rheumatic fever, especially with cardiac localisation or recurrent sore throats.
* Subject with a tendency to develop keloids or hypertrophic scars or any other healing disorders.
* Subject with bleeding, haemostatic disorders.
* Subject having received treatment with a laser, a dermabrasion, a surgery, a chemical peeling or any other procedure based on active dermal response on/around the lips within the past 12 months prior to screening visit or who plans to undergo any of these procedures during the study.
* Subject having received a hyaluronic acid implant into the lips within the past 18 months prior to screening visit or who plans to undergo this procedure during the study.
* Subject having received at any time, any product other than hyaluronic acid into and/or around the lips, like collagen or injection with a slowly resorbable filling product (polylactic acid, calcium hydroxyapatite, combinations of hyaluronic acid (HA) and hypromellose, HA and dextran microbeads or HA and TriCalcium Phosphate (TCP), …) or with a non-resorbable filling product (polyacrylamide, silicone, combination of methacrylic polymers and collagen, polymer particles,...) or who plans to undergo any of these procedures during the study.
* Subject having received at any time a lip threading surgery or who plans to undergo this procedure during the study.
* Subject who received oral surgery (e.g. tooth extraction, orthodontia or implantation) within 6 weeks prior to screening visit or who plans to undergo any of these procedures during the study.
* Subject having started or changed her oral contraceptive or any other hormonal treatment during 12 weeks prior to screening visit.
* Subject using medication such as aspirin, nonsteroidal anti-inflammatory drugs (NSAIDs), antiplatelet agents, thrombolytics, anticoagulants or vitamin C within one week prior to first injection visit (V1) and agreeing not to take such treatments within 1 week prior to touch-up visit (V2) or being a chronic user.
* Subject using medication that reduce or inhibit hepatic metabolism (i.e. protease inhibitors, azole antifungals, macrolides, amiodarone, diltiazem, verapamil, ciprofloxacin, fluvoxamine).
* Total injection volume of cross-linked hyaluronic acid >17,5 mL (whole body) within 1 year prior to screening visit.
* Subject undergoing a topical treatment on the test area or a systemic treatment:

  * Anti-histamines during the 2 weeks prior to injection visit (V1) and agreeing not to take such treatment within 2 weeks prior to touch-up visit (V2);
  * Immunosuppressors and/or corticoids during the 4 weeks prior to screening visit;
  * Retinoids during the 6 months prior to screening visit.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 92 (Actual)
Dates: Start 2021-05-31 (Actual); Primary Completion 2021-10-11 (Actual); Study Completion 2022-07-12 (Actual)

PRIMARY OUTCOMES:
Subject self-assessed global aesthetic evolution of the lips | Month 3
  Proportion of subjects having a positive aesthetic evolution on the 5-point Global Aesthetic Improvement Scale (GAIS) evaluated by the subject on the lips (after mirror self-examination), 3 months after treatment initiation (V1).
  Positive aesthetic evolution according to Global Aesthetic Improvement Scale (GAIS) corresponds to one of these three categories: "Very much improved", "Much improved" or "Improved".
  The 5-point GAIS contains the following categories: "Very much improved", "Much improved", "Improved", "No change" and "Worse".

SECONDARY OUTCOMES:
Subject self-assessed global aesthetic evolution of the lips | Month 1, Month 6, Month 9, Month 12
  Proportion of subjects having a positive aesthetic evolution of the lips at 1, 6, 9 and 12 months, after treatment initiation, as assessed by the subject (after mirror self-examination) using the 5-point Global Aesthetic Improvement Scale (GAIS).
  Positive aesthetic evolution according to Global Aesthetic Improvement Scale (GAIS) corresponds to one of these three categories: "Very much improved", "Much improved" or "Improved".
  The 5-point GAIS contains the following categories: "Very much improved", "Much improved", "Improved", "No change" and "Worse".
Investigator's assessment of global aesthetic evolution of the lips | Month 1, Month 3, Month 6, Month 9, Month 12
  Proportion of subjects having a positive aesthetic evolution of the lips at 1, 3, 6, 9 and 12 months, after treatment initiation, as assessed in live by a blinded independent evaluator using the 5-point Global Aesthetic Improvement Scale (GAIS).
  Positive aesthetic evolution according to Global Aesthetic Improvement Scale (GAIS) corresponds to one of these three categories: "Very much improved", "Much improved" or "Improved".
  The 5-point GAIS contains the following categories: "Very much improved", "Much improved", "Improved", "No change" and "Worse".
Lips' surface aspect | Month 1, Month 3, Month 6, Month 9, Month 12
  Proportion of subjects having a positive aesthetic evolution of the surface aspect of the lips at 1, 3, 6, 9 and 12 months as assessed in live by a blinded independent evaluator using a 5-point questionnaire. For each items of the questionnaire, improvement corresponds to one of these two categories: "Much improved" or "Improved".
  For each of the 5 items of the questionnaire, one of the following answer is selected: "Much improved", "Improved", "No change", "Worsened", "Very worsened"
Evolution of subject's satisfaction | Month 1, Month 3, Month 6, Month 9, Month 12
  Mean changes in subject's satisfaction scores from baseline to 1, 3, 6, 9 and 12 months using the FACE-Q© "satisfaction with lips" questionnaire.
  The FACE-Q© is a patient-reported outcome (PRO) measure of outcomes of aesthetic facial procedures and products from the patient's perspective. The FACE-Q© "satisfaction with lips" is a scale that measures the appearance of the lips with items that ask about size, shape and fullness, as well as how their lips suit their face and how the lips look when smiling.
  For each of the 10 items, one of the following answer is selected: "Very dissatisfied", "Somewhat dissatisfied", "Somewhat satisfied", "Very satisfied".
  Patient responses to each item are graded on a four-point scale and then converted to a score on a scale from 0 (worst) to 100 (best). A higher score means greater satisfaction.
Pain during injection | Day 0, Month 1
  Mean pain scores during injection assessed by the subjects using a 11-point numeric rating scale (0 to 10) at V1 (D0) and V2 (M1) if applicable.
Report of adverse events | Day 0, Month 1, Month 3, Month 6, Month 9, Month 12
  Product tolerance will be assessed by collection of Injection Site Reactions (ISRs) after each injection session, and Adverse Events (AEs) throughout the study. AEs will be summarized by MedDRA System Organ Class and Preferred Term, and will be tabulated by severity, causality, action taken and outcome, using descriptive statistics.

CONTACTS AND LOCATIONS:
Overall Officials: Julia Gotlib, MD, Principal Investigator — Coordinating investigator
Locations (2):
- Eurofins Dermscan Pharmascan, Villeurbanne, France
- Eurofins Dermscan Poland, Gdansk, Poland